CLINICAL TRIAL: NCT04612452
Title: The DTG-SWITCH Study: Longitudinal Analysis of Virologic Failure and Drug Resistance at and After Switching to Dolutegravir-based First-line ART
Acronym: DTG-SWITCH
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: University of KwaZulu (Other); Lighthouse Trust (Other); Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Other Study IDs: DTG-SWITCH Study protocol
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hiv; Drug Resistancy; Virologic Failure
Keywords: Hiv; Drug resistancy; Virologic failure; DTG-based regimen; Drug resistance mutations
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lighthouse Trust in Lilongwe
- CIDRZ in Lusaka

SUMMARY:
This is a prospective observational cohort study of 2820 patients on first-line ART switching to a DTG-based first-line regimen, according to the standard of care. The study is conducted in Malawi and Zambia, in ART programs that participate in the IeDEA collaboration. Sequencing will be done on blood samples of patients with a viral load above 400 copies/mL to identify mutations.

DETAILED DESCRIPTION:
Dolutegravir (DTG), a second-generation integrase strand transfer inhibitor (InSTI), is widely used in high-income countries and is recommended by the World Health Organization (WHO) as an alternative first-line ART regimen. In countries where viral load monitoring is not routinely available many patients on first-line ART will be switched to a DTG-based regimen despite the detectable viral load, which could increase the risk of selection of resistance to DTG as the majority of patients with virologic failure on first-line EFV-based ART have NRTI mutations. The investigators hypothesize that the proportion of patients experiencing virologic failure 48 and 96 weeks after switching to a DTG-based regimen will be higher in patients who switched with virologic failure (VL>400 copies/mL) compared to patients who switched with suppressed viral replication (VL<400 copies/mL). This is a prospective observational cohort study of 2820 patients on first-line ART switching to a DTG-based first-line regimen, according to the standard of care. The study is conducted in Malawi and Zambia, in ART programs that participate in the IeDEA collaboration. At the time of switching to DTG, a baseline study assessment will be done, and a blood sample will be taken. Sequencing will be done on blood samples of patients with a viral load above 400 copies/mL to identify mutations.

ELIGIBILITY:
Inclusion Criteria:

Patients

* On first-line ART for 6 months or longer
* Switching to any DTG-based treatment

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV.
Sampling Method: Non-Probability Sample
Enrollment: 2820 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with VF at 48 weeks between patients with and without VF at baseline. | 48 weeks

SECONDARY OUTCOMES:
The proportion of patients with VF at 96 weeks between patients with and without VF at baseline. | 96 weeks
The incidence of TLD drug resistances at 48 and 96 weeks in patients with and without VF at switch. | 48 and 96 weeks
The proportion of HIV-infected patients with VF at baseline. | Baseline
The proportion of patients with VF at 48 weeks and 96 weeks in patients with VF at baseline who have at least one or no fully active NRTI on resistance testing. | 48 and 96 weeks
Prevalence of neuropsychiatric symptoms at baseline, 48 weeks and 96 weeks. | 48 and 96 weeks
Prevalence of insomnia at baseline, 48 weeks and 96 weeks. | 48 and 96 weeks
Weight change from baseline to 48 and 96 weeks. | 48 and 96 weeks
Levels of adherence at baseline and after 48 and 96 weeks. | 48 and 96 weeks
The number of clinical visits whilst on a DTG-based regimen up to 48 and 96 weeks. | 48 and 96 weeks
The number of clinical visits up to baseline, 48 and 96 weeks. | 48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Egger, Prof., Study Director — University of Berne
Locations (2):
- Lighthouse Trust, Lilongwe, Malawi
- CIDRZ, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Skrivankova VW, Huwa J, Muula G, Chiwaya GD, Banda E, Buleya S, Chihota B, Chintedza J, Bolton C, Tweya H, Kalua T, Hossmann S, Kouyos R, Wandeler G, Egger M, Lessells RJ. Virologic Failure and Drug Resistance After Programmatic Switching to Dolutegravir-based First-line Antiretroviral Therapy in Malawi and Zambia. Clin Infect Dis. 2025 Feb 5;80(1):120-128. doi: 10.1093/cid/ciae261. PMID 38847281